CLINICAL TRIAL: NCT01913847
Title: Phase III Study to Evaluate Efficacy and Safety of HGP1207 in Patients With Pulmonary Hypertension Associated With Systolic Heart Failure
Brief Title: Safety and Efficacy Study of HGP1207 in Patients With Pulmonary Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-SIL-301
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Pulmonary Hypertension; Systolic Dysfunction
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): Sildenafil 20 mg
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Oral sildenafil 20 mg TID for 12 weeks
  Other Names: HGP1207; PAHTENSION chewable tablet
  Arms: Sildenafil
Drug: Placebo — Oral placebo TID for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and clinical efficacy of HGP1207 (Sildenafil) in subjects with pulmonary hypertension associated with systolic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of chronic heart failure (NYHA Class II and III)
* LVEF ≤ 40%
* Elevated systolic PAP: ≥ 40 mmHg
* Patients must be treated with an ACE inhibitor, ARB, beta-blocker, aldosterone antagonist at a stable dose for at least 4 weeks prior to visit 1

Exclusion Criteria:

* Patients with pulmonary hypertension associated with chronic obstructive pulmonary disease, interstitial lung disease, chronic thromboembolism or unclear/multifactorial mechanisms
* Patients who have received Nitrates/NO donor or Cytochrome P450 3A4 inhibitors within 30 days prior to visit 1
* Patients who have received calcium channel blocker, endothelin receptor antagonist, prostacyclin analogues, phosphodiesterase 5 inhibitors within 90 days prior to visit 1
* History of hypersensitivity or allergy to sildenafil or any excipients of its formulation
* Patients with hypertension (sitSBP >170 mmHg or sitDBP>100 mmHg) or hypotension (sitSBP<90 mmHg or sitDBP<50 mmHg)
* Patients with other medical condition (i.e.,alcoholism, drug abuse) that may cause the patient to be non-compliant with the protocol, confound the data interpretation
* Pregnant females or those of child bearing potential who have not had a negative pregnancy test

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 6-min-walk test distance | at 12 weeks

SECONDARY OUTCOMES:
Change from baseline in 6-min-walk test distance | at 6 weeks
Change from baseline in systolic pulmonary arterial pressure (PAP) | at 6 weeks and 12 weeks
Change from baseline in [NT pro-BNP] | at 6 weeks and 12 weeks
Improvement in NYHA functional class | at 6 weeks and 12 weeks
Quality of life (QoL) assessed by EuroQoL(EQ-5D-3L) and EQ visual analogue scales (VAS) | at 6 weeks and 12 weeks
Delaying time to first occurrence of either cardiovascular events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Hyung Ryu, M.D. Ph.D., Principal Investigator — Hallym University Dongtan Sacred Heart Hospital
Locations (1):
- 11 institutions including Hallym University Dongtan Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No